CLINICAL TRIAL: NCT04763174
Title: An mHealth Symptom Management Intervention for Colorectal Cancer Patients
Brief Title: An mHealth Symptom Management Intervention for Colorectal Cancer Patients (mCOPE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107498
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer
Keywords: cancer; pain; fatigue; distress; coping; mHealth; symptom management
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Pain; Fatigue | interventions — Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Coping Skills Training for Symptom Management (mCOPE) (Experimental): mHealth Coping Skills Training for Symptom Management (mCOPE) protocol tests the efficacy of a theory-based symptom management intervention designed to target multiple interrelated symptoms (pain, fatigue, psychological distress) with content uniquely relevant for young and middle-aged colorectal cancer patients. Addressing the co-morbid consequences of cancer while providing support in the context of age-related challenges (e.g., caring for children and parents, career) has the potential to significantly improve overall quality of life in young and middle-aged patients with cancer.
  Interventions: Behavioral: mHealth Coping Skills Training for Symptom Management (mCOPE)
- Standard Care (No Intervention): Standard Care group will complete assessment questionnaires at the same time points as mCOPE, but will not receive mCOPE protocol.

INTERVENTIONS:
Behavioral: mHealth Coping Skills Training for Symptom Management (mCOPE) — mCOPE participants will complete 5 videoconferencing sessions (within 5-9 weeks) with a psychologist, each lasting 45-60 minutes, from a location convenient to the patient (e.g., home, work). Sessions will include cognitive behavioral coping skills designed to target pain, fatigue and psychological distress symptoms unique to colorectal cancer patients. mCOPE will include a mobile app for: 1) coping skills content (e.g., audio, video), 2) daily symptoms assessment and coping skills use tracking transmitting in real-time to study staff, and 4) push notifications for reminders, encouragement, and personalized feedback.
  Arms: mHealth Coping Skills Training for Symptom Management (mCOPE)

SUMMARY:
The investigators have developed an innovative mobile health (mHealth) coping skills training protocol, mCOPE, that is adapted to meet the multiple symptom needs and stage-of-life challenges faced by young and middle-aged adults with cancer, and delivered in a convenient and flexible format that does not incur further demands. Young and middle-aged colorectal cancer patients who report pain, fatigue, and psychological distress will be invited to participate in the study. Participants will be randomly assigned to one of two conditions: mCOPE or standard care. mCOPE will teach patients coping skills to manage their cancer-related symptoms (pain, fatigue and distress) in the context of unique age-related challenges; session content will be tailored based on participants' report. mCOPE sessions will be delivered via videoconferencing to the patient in his/her own environment and scheduled at times that are convenient to the patient. mHealth technology, including a mobile app, will be used to capture daily symptom and coping skills use data, allowing the study team to provide personalized real-time feedback to patients. Investigators want to understand the impact of the mCOPE intervention delivered to young and middle-aged colorectal cancer patients with pain, fatigue, and distress. mCOPE is expected to lead to reduced symptom severity and improved quality of life. Study aims include: testing the efficacy of mCOPE for improving symptoms and quality of life and examining improved self-efficacy for symptom management as a mediator of symptom severity.

DETAILED DESCRIPTION:
There is a high level of evidence that suggests cognitive and behavioral factors play an important role in colorectal cancer patients' abilities to cope with pain, fatigue and distress. Patients with multiple persistent symptoms may be particularly likely to have low confidence in their ability to control their symptoms (i.e., self-efficacy for symptom management). Cognitive behavioral coping skills protocols can enhance patients' abilities to cope with their symptoms in the context of age-related challenges; to date, these protocols have been tested in older patients and neither intervention content nor delivery modality meet the needs of younger patients.

Intervention protocols aimed at young and middle-aged patients dealing with age-related stressors and high time demands must be adapted to meet the needs and challenges (e.g., coping skills practice strategies within the context of competing demands, communication with others about symptoms and limitations, relaxation for managing stoma-related pain, activity pacing to manage fatigue due to cancer and the demands of multiple life roles; cognitive restructuring negative thoughts surrounding managing time off work for treatment while maintaining health insurance and arranging childcare) of younger adults with cancer and delivered in a format (e.g., videoconferencing, adjunctive mobile app) that is acceptable and does not incur further demands.

The investigators propose to use a randomized controlled trial (RCT) to test an innovative mHealth Coping Skills Training for Symptom Management (mCOPE) intervention designed to target pain, fatigue, psychological distress, and quality of life with unique content adapted for young and middle-aged colorectal cancer patients. mCOPE will be delivered with convenient mHealth modalities (videoconferencing, mobile app supported). Young and middle-aged adults with colorectal cancer that endorse multiple symptoms will be randomized to: 1) mCOPE or 2) standard care. mCOPE includes 5 videoconferencing sessions of a cognitive behavior theory-based protocol that teaches coping skills (e.g., relaxation, activity pacing, cognitive restructuring) relevant to managing pain, fatigue and distress, and improving quality of life in the context of the unique challenges facing younger patients. mCOPE uses mHealth technology, including a mobile app, to capture daily symptom and coping skills use data and provide personalized support and feedback to patients. The central hypothesis is that mCOPE will result in decreased pain, fatigue and distress, and increased quality of life.

Specific study aims are:

Aim 1: Test the efficacy of mCOPE for improving symptoms and quality of life.

Aim 2: Examine improved self-efficacy for symptom management as a mediator of symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of colorectal cancer within the past three years
* Stages I-IV
* Reported pain, fatigue and psychological distress - minimum two of three symptoms reported at 3 or greater on 0-10 scale
* Able to speak and read English

Exclusion Criteria:

* Cognitive impairment (e.g., dementia)
* Presence of a severe psychiatric condition (i.e., psychotic disorder or episode) or a psychiatric condition (e.g., suicidal intent)
* Participation in a coping skills training protocol in the past 6 months
* Inability to converse in English

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 167 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Change in pain severity | Baseline, post-intervention (up to 10 weeks post-intervention), 3-month, and 6-month: approximately 20 minutes each time.
  Pain Severity will be assessed using the Brief Pain Inventory (BPI) by asking patients about worst, least, average and now pain on a 0 = no pain to 10 = pain as bad as you can imagine.
Change in fatigue | Baseline, post-intervention (up to 10 weeks post-intervention), 3-month, and 6-month: approximately 20 minutes each time.
  The Patient Reported Outcomes Measurement Information System (PROMIS) seven-item Fatigue Scale is a self-report measure of fatigue symptoms. Items ask patients to evaluate symptoms from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that is likely to decrease one's ability to carry out daily activities.
Change in psychological distress | Baseline, post-intervention (up to 10 weeks post-intervention), 3-month, and 6-month: approximately 20 minutes each time.
  The Brief Symptom Inventory (BSI) will be used to measure psychological distress. Responses are rated on a 5-point scale where 0=not at all and 4=extremely for questions such as "feeling not interested in things" and "feeling hopeless about the future."

SECONDARY OUTCOMES:
Change in quality of life | Baseline, post-intervention (up to 10 weeks post-intervention), 3-month, and 6-month: approximately 20 minutes each time.
  The Functional Assessment of Cancer Therapy - General (FACT-G), version 4.0, is a 27-item self-report measure that assesses quality of life concerns specific to cancer patients. FACT-G is comprised of four quality of life domains including physical, social/family, emotional, and functional well-being.
Change in Self-Efficacy for Symptom Management | Baseline, post-intervention (up to 10 weeks post-intervention), 3-month, and 6-month: approximately 20 minutes each time.
  Self-Efficacy for Symptom Management will be assessed using the Patient Reported

OTHER OUTCOMES:
Change in Psychological Services | Baseline, post-intervention (up to 10 weeks post-intervention), 3-month, and 6-month: approximately 20 minutes each time.
  One item will be asked at each assessment time-point to assess participants' use of psychological services during the course of the study.
Change in Parenting Concerns | Baseline, post-intervention (up to 10 weeks post-intervention), 3-month, and 6-month: approximately 20 minutes each time.
  Parenting Concerns Questionnaire (PCQ) asks in the past month, to what extent have you been concerned with a list of parenting concerns from 1 (not at all concerned) to 5 (extremely concerned). The higher the score, the more concerned.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Kelleher, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Regional Hospital, Durham, North Carolina
  - Duke Cancer Institute, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No